CLINICAL TRIAL: NCT04769622
Title: Influence of Environmental Factors on the Efficacy of Non-surgical Periodontal Treatment. A Pre-post Quasi-experimental Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Researcher, University of Siena
Other Study IDs: NST001
Record Dates: First submitted 2021-02-16; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non Surgical Periodontal Treatment; Periodontitis; Periodontal Diseases
Keywords: periodontitis; non surgical periodontal treatment
MeSH Terms: conditions — Periodontitis; Periodontal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients affected by untreated Periodontitis: patients coming to the Unit of Periodontics at the University of Siena will be screened for the inclusion in the study. All patients eligible for the inclusion in the study will undergo non-surgical periodontal treatment and will be administered a questionnaire about lifestyles (adherence to mediterranean diet, sleep quality, physical activity, perceived stress). Patients will be then reevaluated at 3 months after the completion on non-surgical periodontal therapy.
  Interventions: Procedure: Non-surgical periodontal treatment; Other: Questionnaires

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — all included patients will be subjected to non-surgical periodontal therapy
Other: Questionnaires — All patients will be asked to complete a set of questionnaires regarding:
  * adherence to Mediterranean Diet;
  * sleep quality;
  * physical activity;
  * perceived stress.

SUMMARY:
Periodontitis is a biofilm-mediated chronic inflammatory disease which causes the destruction of the supporting tissues of the tooth. Risk factors for periodontitis include familiarity for periodontal diseases, diabetes, cardiovascular diseases, metabolic syndrome, obesity and stress. Some studies demonstrated how these risk factors negatively influence the patients' response to non-surgical periodontal treatment. The success of non-surgical periodontal therapy is defined through the treat-to-target concept (i.e. a maximum of 4 sites with Probing Pocket Depth >5mm and presence of Bleeding on Probing); therefore, periodontal treatment is successful whenever this threshold is reached. Moreover, given the available data regarding the association between more severe forms of periodontitis and a lower frequency of physical activity, a worse sleep quality and more perceived stress, it is reasonable to hypothesize that these factors could influence the patients' response to non-surgical periodontal treatment. With regards to diet, despite many studies appraised the anti-inflammatory effect of the mediterranean diet, no study has ever related adherence to Mediterranean Diet to oral health status. The novelty that the present study would introduce is the evaluation of how environmental factors (i.e. diet, physical exercise, perceived stress) influence patients' response to non-surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old;
* presence of untreated periodontitis (Papapanou at al. 2018);
* ability and willingness to give informed consent.

Exclusion Criteria:

* pregnancy or lactation;
* patients who underwent non-surgical periodontal therapy in the last 6 months;
* patients taking immunosuppressive drugs;
* inability or unwillingness to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with untreated periodontitis coming to the Unit of Periodontics at the University of Siena and meeting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
Treat-to-target after treatment (yes/no) | outcome measured at reevaluation (3 months after the completion of non-surgical periodontal treatment)
  Binary outcome defining the success of non-surgical periodontal treatment. The treat-to-target is reached whenever patients at reevaluation have a maximum of 4 sites with Probing Pocket Depth (PPD) >5mm and presence of Bleeding on Probing (BoP)

SECONDARY OUTCOMES:
Influence of adherence to Mediterranean diet on the success of non-surgical periodontal treatment (treat-to-target) | outcome measured at reevaluation (3 months after the completion of non-surgical periodontal treatment)
  results obtained from the questionnaire about adherence to Mediterranean Diet (Gnagnarella et al. 2018) will be placed in a logistic regression model, whose aim will be to investigate the influence of adherence to Mediterranean diet (predictors) on the success of non surgical periodontal treatment (treat to target; dependent variable). Adherence to Mediterranean diet is evaluated on a scale between 0 and 9; the higher the score, the higher the adherence to Mediterranean Diet.
Influence of Sleep Quality on the success of non-surgical periodontal treatment (treat-to-target) | outcome measured at reevaluation (3 months after the completion of non-surgical periodontal treatment)
  results obtained from the questionnaire about Sleep Quality (Pittsburgh Sleep Quality Index) will be placed in a logistic regression model, whose aim will be to investigate the influence of sleep quality (predictor) on the success of non surgical periodontal treatment (treat to target; dependent variable). Sleep quality is evaluated on a scale between 0 and 21; the higher the score, the poorer the Sleep Quality.
Influence of Physical Activity on the success of non-surgical periodontal treatment (treat-to-target) | outcome measured at reevaluation (3 months after the completion of non-surgical periodontal treatment)
  results obtained from the questionnaire about Physical Activity (International Physical Activity Questionnaire) will be placed in a logistic regression model, whose aim will be to investigate the influence of amount of Physical activity (predictor) on the success of non surgical periodontal treatment (treat to target; dependent variable). Physical activity is evaluated on a scale between 0 and 2 (0= low physical activity; 1= moderate physical activity; 2= intense physical activity).
Influence of Perceived Stress on the success of non-surgical periodontal treatment (treat-to-target) | outcome measured at reevaluation (3 months after the completion of non-surgical periodontal treatment)
  results obtained from the questionnaire about Perceived stress (Italian Perceived Stress Scale) will be placed in a logistic regression model, whose aim will be to investigate the influence of perceived stress (predictor) on the success of non surgical periodontal treatment (treat to target; dependent variable). Perceived Stress is evaluated on a scale between 0 and 40; the higher the score, the higher the stress perceived.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy